CLINICAL TRIAL: NCT00290017
Title: A Phase 3, Randomized, Double-Blind, Multicenter Study of Talabostat and Pemetrexed vs. Pemetrexed and Placebo in Patients With Advanced (Stage IIIB/IV) Non-Small Cell Lung Cancer (NSCLC) After Failure of Platinum-Based Chemotherapy
Brief Title: Study of Talabostat and Pemetrexed vs. Pemetrexed in Stage IIIB/IV Non-Small Cell Lung Cancer (NSCLC) After Failure of Platinum-Based Chemotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA Hold May 2007
Sponsor: Point Therapeutics (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PTH-305
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Cancer; Neoplasms, Lung; Neoplasms, Pulmonary
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — talabostat; Pemetrexed

INTERVENTIONS:
Drug: talabostat
Drug: pemetrexed

SUMMARY:
This Phase 3 study will compare the efficacy of talabostat plus pemetrexed to pemetrexed plus placebo in patients with Stage IIIB/IV NSCLC who have failed a platinum-based chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age ≥18 years
* Histologically or cytologically confirmed NSCLC (Recurrent, locally advanced or metastatic, inoperable NSCLC [Stage IIIB/IV]. Patients with Stage IIIB NSCLC must have a cytologically documented pleural effusion.)
* Failed or relapsed after receiving a platinum-containing chemotherapy regimen as first-line therapy for advanced NSCLC
* Measurable disease on computerized tomography (CT) scan
* ECOG Performance Status of 0 or 1
* Expected survival ≥12 weeks
* Provide written informed consent

Exclusion Criteria:

* More than 2 prior chemotherapy regimens
* Progression of disease on prior pemetrexed treatment
* Brain metastases (exception: patients who had a resection and/or completed a course of cranial irradiation, have no worsening CNS symptoms, and have discontinued all corticosteroids for that indication for at least 1 month)
* Serum creatinine ≥2.0mg/dL or creatinine clearance <45mL/min
* Absolute neutrophil count <1500/μL or platelets <100,000/μL
* Any malignancy within 5 years immediately prior to the first dose of study medication (exception: basal cell or non-metastatic squamous cell carcinoma of the skin, and carcinoma in-situ of the cervix)
* Any comorbidity or condition which, in the opinion of the investigator, may interfere with the assessments and procedures of this protocol
* Patients who are within 28 days of chemotherapy, radiation therapy, immunotherapy, or investigational medication for NSCLC. Patients must have recovered from all of the side effects of treatment.
* Pregnancy or lactation. Women of childbearing potential and non-vasectomized men must agree to use a barrier method of contraception during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-02

CONTACTS AND LOCATIONS:
Locations (101):
- United States (101):
  - Marshall Schreeder, MD, Huntsville, Alabama
  - Hematology Oncology Associates, Phoenix, Arizona
  - Heritage Physician Group-Oncology, Hot Springs, Arkansas
  - Raul R. Mena, MD, Burbank, California
  - Pacific Coast Hematology / Oncology Medical Group, Inc., Fountain Valley, California
  - Robert A. Moss, MD, FACP, Inc., Fountain Valley, California
  - Antelope Valley Cancer Center, Lancaster, California
  - Warren Paroly, MD, Oceanside, California
  - Southwest Cancer Care Medical Group, Poway, California
  - Mile High Oncology, Denver, Colorado
  - Medical Specialists of Fairfield, Fairfield, Connecticut
  - Northwestern Connecticut Oncology Hematology Associates, LLP, Torrington, Connecticut
  - Lucio Gordan, MD, Gainesville, Florida
  - Cancer and Blood Disease Center, Lecanto, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Center of Florida, Ocoee, Florida
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Hematology Oncology Associates of Illinois, Chicago, Illinois
  - Joliet Oncology-Hematology Associates, Joliet, Illinois
  - American Health Network of Indiana--Hematology/Oncology, Indianapolis, Indiana
  - Arnett Cancer Center, Lafayette, Indiana
  - Northern Indiana Oncology Associates, South Bend, Indiana
  - Associated Physicians and Surgeons, LLC, Terre Haute, Indiana
  - HUX Cancer Center/Union Hospital, Terre Haute, Indiana
  - Kansas City Cancer Center, LLC, Overland Park, Kansas
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Mercy Medical Center, Baltimore, Maryland
  - Chesapeake Oncology Hematology Associates (Tate Center), Glen Burnie, Maryland
  - Carroll County Cancer Center, Westminster, Maryland
  - Fallon Clinic, Inc. at Worcester Medical Center, Worcester, Massachusetts
  - Michael McKenzie, DO, Clinton Township, Michigan
  - Youssef Hanna, MD, Port Huron, Michigan
  - Cancer and Transplant Consultants, PLC, Rochester Hills, Michigan
  - Cancer Care Associates, Rochester Hills, Michigan
  - Cancer Care Associates, PC, Royal Oak, Michigan
  - Hematology Oncology Consultants, Royal Oak, Michigan
  - Jeffrey H. Margolis, MD, Royal Oak, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Dr. Folbe, MD/PC, Troy, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - Minnesota Oncology Hematology, PA, Burnsville, Minnesota
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Hematology Oncology Associates, SJ, PA, Mount Holly, New Jersey
  - Capital Health System, Trenton, New Jersey
  - Mercer Bucks Oncology/Hematology, Trenton, New Jersey
  - New York Oncology Hematology, PC, Albany, New York
  - Northwestern Carolina Oncology & Hematology, PA, Hickory, North Carolina
  - Eugene Paschold, MD, Winston-Salem, North Carolina
  - Piedmont Hematology Oncology / Winston-Salem, Winston-Salem, North Carolina
  - Oncology/Hematology Care, Inc., Cincinnati, Ohio
  - Dayton Oncology & Hematology, PA, Kettering, Ohio
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Satish A. Shah, MD, Gettysburg, Pennsylvania
  - Medical Oncology Associates of Wyoming Valley, PC, Kingston, Pennsylvania
  - Hematology-Oncology Group, PC, Langhorne, Pennsylvania
  - St. Mary Medical Center--Research Center, Langhorne, Pennsylvania
  - Paoli Hospital, Paoli, Pennsylvania
  - Rittenhouse Hematology Oncology Associates, Philadelphia, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Bux-Mont Oncology-Hematology, Sellersville, Pennsylvania
  - Grandview Hospital, Sellersville, Pennsylvania
  - Cancer Care Institute of Carolina, Aiken, South Carolina
  - Charleston Hematology Oncology, PA, Charleston, South Carolina
  - Palmetto Hematology Oncology PC, Spartanburg, South Carolina
  - Associates in Oncology and Hematology, Chattanooga, Tennessee
  - McLeod Cancer and Blood Center, Johnson City, Tennessee
  - University of Tennessee, Knoxville, Tennessee
  - Texas Cancer Center, Arlington, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - Texas Cancer Center (Dallas Southwest), Dallas, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Texas Cancer Center / Denton, Denton, Texas
  - El Paso Cancer Treatment Center--East, El Paso, Texas
  - Texas Oncology, PA, El Paso, Texas
  - Texas Oncology, PA, Fort Worth, Texas
  - US Oncology Research and Clinical Pharmacy, Fort Worth, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Texas Oncology, PA, Mesquite, Texas
  - Texas Oncology, PA / Allison Cancer Center, Midland, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - Texas Oncology Cancer Center--Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Cancer Outreach Associates, PC / Outreach Clinical Trial Consortium LLC, Abingdon, Virginia
  - Fairfax Northern Virginia Hematology / Oncology, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Physicians, Inc., Richmond, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Salem, Virginia
  - Luke Walker, MD, Everett, Washington
  - Cascade Cancer Center, Kirkland, Washington
  - Puget Sound Cancer Centers, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Northwest Cancer Specialists, PC, Vancouver, Washington
  - Medical Consultants, Ltd., Milwaukee, Wisconsin